CLINICAL TRIAL: NCT05041959
Title: Nicotine Withdrawal and Reward Processing
Acronym: NicWith
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: Oklahoma State University (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: K23DA042898 (NIH); K23DA042898 (NIH)
Record Dates: First submitted 2021-09-03; First posted 2021-09-13 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Cigarette Smoking; Nicotine Dependence; Nicotine Withdrawal
MeSH Terms: conditions — Cigarette Smoking; Tobacco Use Disorder

STUDY DESIGN:
Intervention Model Description: Participants will abstain from smoking for 24 hours before one MRI scan and continue smoking as usual before the other
Masking Description: This is a smoking abstinence manipulation. No masking is possible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smoking Abstinence (Other): Participants will abstain from smoking for 24 hours before one MRI scan. Smoking abstinence will be confirmed using exhaled carbon monoxide breath testing
  Interventions: Other: Smoking Abstinence
- Ad Lib Smoking (Other): Participants will continue smoking as usual (i.e. "ad lib") before one MRI scan and smoke one additional cigarette immediately prior to scanning. Continued smoking will be confirmed using exhaled carbon monoxide breath testing.
  Interventions: Other: Ad Lib Smoking

INTERVENTIONS:
Other: Smoking Abstinence — Participants will abstain from smoking for 24 hours
  Arms: Smoking Abstinence
Other: Ad Lib Smoking — Participants will continue smoking as usual (i.e. ad lib) in the day leading up to the scan and smoke one cigarette of their own brand immediately prior to scanning.
  Arms: Ad Lib Smoking

SUMMARY:
This study is designed to find out how smoking affects the way the brain responds to pleasure and how this impacts smokers' behavior. Participants will complete three sessions. The first session will be a screening and training visit to determine final eligibility. Eligible participants will work with a researcher to develop brief scripts about times when they smoke and do other activities. Next, participants will attend two magnetic resonance imaging (MRI) scans - one after abstaining from smoking for 24 hours and the other after smoking as usual. After the second MRI, participants will answer questions on their phone every day for two weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Generally healthy
2. Age 21-55
3. Right-handed using a three-item scale
4. Daily smoker of ≥ 6 cigarettes/day
5. Smoking regularly for ≥ 1 year
6. Have a smartphone capable of running the MetricWire application
7. Able to read and understand English
8. Able to identify at least 6 pleasurable activities they do not do concurrently with smoking or associate with smoking.
9. Able to identify at least 6 unique locations/scenarios they do associate with smoking

Exclusion Criteria:

1. Planning to quit smoking within the next 60 days
2. Currently seeking or receiving treatment for smoking cessation
3. Use of smokeless tobacco, nicotine replacement products or electronic cigarettes more than 5 days in the past month.
4. Breath alcohol level ≥.001. Participants may be allowed one reschedule at the discretion of the PI or other study staff.
5. Positive toxicology screen for illicit drugs

   1. Marijuana will be tested for but will not be exclusionary
   2. Participants failing the toxicology screen may be allowed one re-screening attempt at the PI's discretion
   3. Participants with valid prescriptions who report using the medication as directed and meet all other eligibility criteria may be allowed to participate at the PI's discretion
6. Current use of antipsychotic or stimulant medications.
7. Significant health problems or those that would impact scientific goals of the project, including (but not limited to):

   1. Cancer, Bronchitis, Emphysema, COPD
   2. Asthma or Breathing Problems
   3. Insulin-Dependent Diabetes
   4. Heart disease, angina, heart failure, serious arrhythmia or heart attack within the past 6 months
   5. Systolic Blood Pressure > 160, Diastolic Blood Pressure > 100, HR > 115 bpm (one re-screen allowed).
   6. Glaucoma, color blindness or an uncorrected vision problem
   7. Significant hearing loss requiring the use of hearing aids or other hearing problems that would impact
   8. History of stroke, brain tumor, seizure disorder, or traumatic brain injury
   9. Metal implants (e.g. pacemaker, surgical pins, certain dental repairs), dental braces, or metal fragment injuries.
   10. Claustrophobia
   11. Weight > 350 pounds or unable to fit in the MRI scanner bore
   12. Current psychotic disorder, alcohol use disorder or drug use disorder for drugs other than cannabis (moderate or severe only, mild is allowable at PI's discretion). AUD and DUD in remission are also allowable at PI's discretion.
   13. Pregnant, breastfeeding or planning to become pregnant during the course of the study (females)
8. Current enrollment in another smoking research study or having participated in a study involving daily use of Spectrum cigarettes or other reduced nicotine products within the past three months
9. Irregular sleep-wake cycles (e.g. swing-shift work, unusual sleep pattern)

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2022-06-02 (Actual); Primary Completion 2024-03-29 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
Blood Oxygen Level Dependent (BOLD) Activation | Approximately 2-4 weeks
  BOLD activation in brain reward network regions
Ecological Momentary Assessment (EMA) Pleasure Ratings | 2-4 weeks
  Anticipated and experienced pleasure based on self-report ratings acquired each day during the EMA phase

CONTACTS AND LOCATIONS:
Locations (1):
- Hardesty Center for Clinical Research and Neuroscience, Tulsa, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: Yes
Detailed protocols, datasets and additional information will be available from the Principal Investigator and research team upon request. In order to maintain compliance with the Health Insurance Portability and Accountability Act (HIPAA) requirements, as well as university data security policies, all data will be anonymized according to HIPAA guidelines prior to being shared. Individual participant scripts will not be made publicly available due to privacy concerns and because this could impact the nature of information participants were willing to provide for scripts. Data will be provided in widely accessible formats for both self-report and imaging data. We will work with relevant administrative offices to obtain guidance regarding any required Data Use Agreements as needed.
Supporting Information: Study Protocol
Time Frame: We anticipate making data available within 6 months of study completion. It will be available for an indefinite period of time.
Access Criteria: Contact PI for details.